CLINICAL TRIAL: NCT01154595
Title: Effectiveness and Cost-effectiveness of a Ready-to-Use-Food (RUF) Supplement to Prevent Acute Malnutrition in Children Between 6-36 Months in Urban Chad
Brief Title: Effectiveness of a Ready-to-Use-Food (RUF) Supplement to Prevent Acute Child Malnutrition
Acronym: PREAMA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Action Contre la Faim (Other)
Collaborators: University Ghent (Other)
Responsible Party: Principal Investigator, Lieven Huybregts, Principal Investigator, University Ghent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UGENT0410
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Child; Malnutrition
Keywords: moderate acute malnutrition, prevention, Lipid-based supplement
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Food-for-Training component (Active Comparator): Conditional family food supplementation (sugar, sorghum, beans, iodized salt, vegetable oil) 1800 kcal/person/day in function of attendance and participation in a sensitization program covering various themes on household, water and disease management, hygiene promotion, sanitation and dietary practices for children.
  Interventions: Behavioral: Food-for-Training
- Food-for-Training + RUF (Plumpy Doz(r)) (Experimental): Conditional family food supplementation (sugar, sorghum, beans, iodized salt, vegetable oil) 1800 kcal/person/day in function of attendance and participation in a sensitization program covering various themes on household, water and disease management, hygiene promotion, sanitation and dietary practices for children.
  In addition, a blanket supplementation with 47g RUF (Plumpy Doz(r)) per day per child is provided.
  Interventions: Dietary Supplement: Plumpy Doz(r) - Ready-to-Use Food; Behavioral: Food-for-Training

INTERVENTIONS:
Dietary Supplement: Plumpy Doz(r) - Ready-to-Use Food — 47g Plumpy Doz(r) per day per child
  Arms: Food-for-Training + RUF (Plumpy Doz(r))
Behavioral: Food-for-Training — Conditional family food supplementation (sugar, sorghum, beans, iodized salt, vegetable oil) 1800 kcal/person/day in function of attendance and participation in a sensitization program covering various themes on household, water and disease management, hygiene promotion, sanitation and dietary practices for children.

SUMMARY:
The overall objective of this project is to assess the effectiveness and cost-effectiveness of RUF (ready-to-Use Food, Plumpy Doz(r)) to prevent moderate acute malnutrition in children aged 6-36 months if embedded in a program of conditional household food assistance.

ELIGIBILITY:
Inclusion Criteria:

* WH≥80% of median of NCHS reference without bilateral pitting oedema;
* Age ≥ 6 months and ≤36 months;
* Member of a household with a dependency ratio >4;
* Not planning to leave the study zone for the coming 5 months;

Exclusion Criteria:

* Not showing appetite;
* Age < 6 months or age > 36 months
* Weight-for-Height Z-score <-2 and/or the presence of bilateral pitting oedema in children 6-36 months;
* Member of a household with a dependency ration ≤ 4;
* Clinical complications
* Presence of chronic illness, cardiac disease, congenital abnormalities, cancer;
* Being allergic to one of the ingredients of the RUF.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Cumulative wasting incidence, hemoglobin concentration | monthly

SECONDARY OUTCOMES:
weight gain | monthly
time to become wasted | monthly
default rate | monthly
RUF acceptability | monthly
dietary intake | monthly

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Kolsteren, PhD MD, Principal Investigator — University Ghent; Lieven Huybregts, PhD, Principal Investigator — University Ghent
Locations (1):
- Action Contre La Faim Tchad, Abéché, Chad

REFERENCES:
- [Derived] Huybregts L, Houngbe F, Salpeteur C, Brown R, Roberfroid D, Ait-Aissa M, Kolsteren P. The effect of adding ready-to-use supplementary food to a general food distribution on child nutritional status and morbidity: a cluster-randomized controlled trial. PLoS Med. 2012;9(9):e1001313. doi: 10.1371/journal.pmed.1001313. Epub 2012 Sep 18. PMID 23028263